CLINICAL TRIAL: NCT06766409
Title: The Effectiveness of Joint Provision of Community Group-based Family Planning Counseling with Routine Individual Counseling Provided to Perinatal Women on Postpartum Contraception Acceptance
Brief Title: Effect of Joint Provision of Community Group-based Counseling with Individual Counseling on Postpartum Contraception
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Paul's Hospital Millennium Medical College, Ethiopia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Stpaulhospitalmilleniummedical
Record Dates: First submitted 2024-12-25; First posted 2025-01-09 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-12

CONDITIONS: Postpartum Contraception
Keywords: Postpartum contraception; Postpartum family planning; Ethiopia

STUDY DESIGN:
Intervention Model Description: A two-arm parallel cluster randomized control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group-based counseling (Active Comparator): A perinatal woman in the intervention arm will receive group-based family planning counseling at the community level, which includes a process of arranged demonstration of all available family planning methods jointly with routine individual family planning counseling.
  Interventions: Behavioral: A community group-based demonstration counseling method
- Individual-based counseling (Placebo Comparator): Prenatal and postnatal women in the control arm will just receive routine individual FP counseling only based on the Ethiopian national guidelines.
  Interventions: Behavioral: An individual family planning counseling

INTERVENTIONS:
Behavioral: A community group-based demonstration counseling method — At the community level, a perinatal woman in the intervention arm will get individual family planning counseling along with group-based counseling that includes a planned demonstration of all possible techniques.
  Arms: Group-based counseling
Behavioral: An individual family planning counseling — The control group's pregnant and postpartum women will simply get standard individual FP counseling in accordance with Ethiopian national recommendations.
  Arms: Individual-based counseling

SUMMARY:
The aim of this trial is to assess the effectiveness of joint provision of community group-based demonstration counseling methods with routine individual family planning counseling provided to prenatal and postnatal women on postpartum contraception acceptance in the West Shoa Zone, Oromia, Ethiopia. A two-arm cluster randomized control trial will be conducted to compare the routine individual facility-based family planning counseling with the joint provision of individual and community group-based counseling with a process of arranged demonstration on the later part. The study will be conducted from March 1, 2025, to May 30, 2026. A sample of 598 women (21 women per 28 clusters) will be selected by a two-stage (stratification and clustering) sampling. A structured questionnaire will be used to collect the data. The data will be entered into STATA (V16). A goodness of fit test using Pearson's chi-square and a multicollinearity test will be checked. Multinomial logistic regression will be used for analysis.

The main questions it aims to answer are:

1. Will postpartum women in the intervention group (joint provision of individual and community group-based counseling) be more likely to use contraception?

   1. Percent of postnatal women who receive any method from the intervention group.
   2. Percent of postnatal women who receive any method from the control group.
2. Will postpartum women in the intervention group, subject to an intervention group, prefer highly effective contraceptive methods?

   1. Percent of postnatal women who receive highly effective methods from the intervention group.
   2. Percent of postnatal women who receive low-effective methods from the control group.
   3. Percent of postnatal women who receive highly effective methods from the control group.
   4. Percent of postnatal women who receive low-effective methods from the intervention group.

DETAILED DESCRIPTION:
Introduction

World Health Organizations recommend postpartum family planning as a critical component of health care that has the potential to meet women's desire for contraception and save millions of maternal and infant lives in low- and middle-income countries. It recommends that after "a woman gave birth," she should avoid pregnancy for at least two years prior to the next pregnancy to ease the maternal, prenatal, and infant risks. It is also an important determinant of women's ability to exercise their reproductive autonomy and a key facilitator of gender equality and women's empowerment. Additionally, it is a key to achieving global public health goals, such as the Sustainable Development Goals on sexual and reproductive health.

Therefore, it is crucial to start using contraception as soon as possible after giving birth because it lowers the risk of an unwanted pregnancy and prolongs the time between pregnancies, which benefits both mothers and newborns' health. Contraceptive plans should optimally be initiated as part of prenatal care and counseling, especially as many methods can be provided at the time of delivery or during the hospital stay. When contraceptive counseling is offered during both the prenatal and postpartum periods, the prevalence of postpartum contraceptive use, including the use of more effective methods, is highest, especially when it is offered in group-based compared to individual counseling. Maternal and infant mortality can be prevented by combining prenatal care, family planning, postpartum care, vaccination, and nutrition programs as an integrated service.

Methods

This study is designed as a two-arm, unblinded, cluster randomized controlled trial with baseline and follow-up measurements. Perinatal women among the study participants will be randomly assigned to each arm. One arm includes routine individual family planning counseling only, and the other group includes joint provision of community group-based counseling with routine individual counseling. The trial protocol will be developed, delivered, and reported in accordance with the Consolidated Standards of Reporting Trials (CONSORT) guidelines. The study participants will be women with near-term, term, and post-term pregnancies and postnatal women who live in the West Shoa Zone.

A community-group-based counseling program, which includes a process of arranged demonstration of all available methods, will be provided to women with a prenatal period beyond 34 completed weeks of pregnancy and postnatal women in the intervention group. The purpose of the demonstration method will be to improve the recall status, decision-making ability, and informed free choice of postnatal women on contraception. The arranged demonstration method will be prepared with all available contraceptive methods, posters, and other visual aids. The expert in this area will arrange a community-based demonstration counseling method step-by-step for 30 minutes that creates free discussion and a flow of opinions among the participants. Participants can find real-time information about contraceptive methods, including the advantages, side effects, how they receive them, for how long, if there is any cost for the methods, and if there is any indication to discontinue or change the method. A facilitator's guide will provide step-by-step details on how to conduct a demonstration. The guided discussions on family planning will be provided based on World Health Organization guidelines and communication tools. They are structured on the basis of social cognitive theory, addressing factors that could help reduce risk-taking and improve self-efficacy and motivation, and in motivational interviewing, with active listening and a non-judgmental attitude. The group counseling will be provided at the community setting (Kebeles and school sites). Both groups will complete a first questionnaire at baseline (T0) and at the endline (12 months after T0). The time will be chosen to coincide with the dates of their postpartum care and immunization schedules. Because at this time is also one of the contact points for family planning integration with other services, and most women schedule for family planning during immunization periods. Participants will be given the leaflet and other visual aids as an incentive. In general, a significant change in the use of and preferences for contraceptive methods among postnatal women in the control group will not be expected compared to those women who receive both individual and group-based counseling. In Ethiopia, the study also revealed some weaknesses in the trends of routine family planning counseling.

The sample size will be calculated to detect a 15-percentage-point difference in postpartum contraception between the two arms. The baseline prevalence of postpartum contraception was estimated to be 40% in Ethiopia, based on the most recent Demographic and Health Survey (DHS) estimates. The assumptions include an intra-cluster correlation coefficient (ρ = 0.03) (based on the previous similar study), an expected rate of 55% of intervention group women and 40% of control group women showing postpartum contraceptive use (a primary outcome), with an alpha level of 0.05 after 1 year from baseline. The assumptions also include a 95% confidence interval (CI), 10% non-response, design effect, or so-called variance inflation factor (1+ρ(m-1)) (1+ 0.03 (21-1) of cluster design of 1.6), and a sample size ratio of 1 between the control and intervention groups. Statistical power will be individually maximized after considering sample-size constraints, including the estimated number of eligible clusters. The resulting power is 80% with a final sample calculation of 299 post-natal women in each arm (598 sample women for both groups).

A cluster in this study is defined as the residence of prenatal and postnatal women who meet inclusion criteria. The reasoning behind randomizing clusters rather than individual women is that women residing in the same residence will likely have more similar experiences than those living in different residences. In the hypothetical case where randomization is performed at the individual level, then individual women in the same residence could be randomized to different intervention groups. If so, there would be a greater likelihood of statistical 'contamination' whereby women within a residence in the intervention group might share information from the arranged demonstration method with those assigned to the control group within the same residence. The cluster randomized control trial helps to avoid this potential for contamination. Random assignment of clusters to intervention or control groups will use a 1:1 randomization ratio without restriction (completely randomized). Therefore, random sampling will be done in two stages. In the first stage, randomization will be stratified by the woman's residence. There are 584 kebeles in the West Shoa Zone Oromia Region, and they will be stratified into two strata (stratum 1 = 55 urban kebeles and stratum 2 = 529 rural kebeles) based on geographical location. Each kebele is considered a cluster. The unit of randomization in this step is a cluster (kebele). Then, using the simple random sampling technique, 14 kebele will be randomly selected to be the intervention kebele, and 14 kebele will be selected to be the control kebele, for a total of 28 kebeles. After then, all pregnant (late) and postpartum women in the chosen cluster will be enrolled for the 12-month postpartum period. Approximately two weeks before recruitment, first conduct a door-to-door household enumeration will be conducted to identify study-eligible women among the selected clusters (kebeles).

Recruitment and data collection will be from March 2025 to March 2026. A trained health provider will employ a structured questionnaire. The study will enroll women in three phases to fit their pregnancy and postnatal schedules. The participants will be divided into different cohorts and receive the intervention separately. The first cohort of women includes prenatal women in their late pregnancy (near term, term, and post-term). Those cohorts will receive the intervention 3 times: before delivery (T0), at six months (T1), and nine months (T2) postpartum. The second cohort will be postnatal women with less than 6 months. Those groups will receive the intervention 2x: at six months (T0) and 9 months (T1) postpartum. The third cohort will be women whose postpartum period is between six and nine months. Those will receive the intervention at nine months. All cohorts will receive and fill the baseline questionnaire at the beginning of the study (T0) and the endline questionnaire at 12 months (1 year) post-delivery. The baseline questionnaire will be completed at T0. After the baseline questionnaire, the clusters/Kebeles will be randomly assigned to one of the two intervention arms: routine family planning counseling only or joint provision of routine individual counseling and group-based. During the community house screening, all selected women will be contacted at community settings.

The questionnaire that will be used for this study is adopted from a pre-validated questionnaire that has been used for studies on the same area of research questions. It will also be guided by Ethiopian national guidelines for family planning services. Similar questions to those found in Demographic and Health Surveys are included in the questionnaire. The use of methods will be assessed by asking which form or forms of contraception (if any) they are currently using and how these methods will be used. The questionnaire will be administered by trained midwives in both groups. A structured questionnaire will be prepared in English, translated to A/Oromo, and then back to English by a professional translator to check for consistency of the questions and comparability of the findings. The translation will be done to meet the understanding of local participants with the Amharic and A/Oromo tongues. Moreover, experts will review the content validity of the questionnaires, which will be followed by a pre-test to identify changes and clarify any ambiguity. Pre-tests of the data collection tools will be conducted with 5% of the sample size from a population with similar characteristics. Once this pre-test data has been analyzed, the required adjustments will be made prior to data collection. The collected data will be checked for completeness and inconsistencies before data processing. Participants who do agree to participate will be asked to provide written informed consent. The project will collect comprehensive baseline data on women's demographics, socio-economic status, medical history, reproductive history, and past and current pregnancy-related factors. During the baseline and endline questionnaire, the women will be assessed for contraceptive use and method choices.

The baseline data that will be collected from the study participants will be entered into a Kobo toolbox, and the data will be cleaned and exported to STATA version 16. Changes in the primary outcome will be analyzed by using data from the full-analysis set, which included all participants who underwent randomization (intention to treat). The adjusted odds ratio will be reported as the baseline parameter using postpartum contraceptive use as an outcome variable while adjusting for age, type of family, marital status, education, family income, occupation, number of successful deliveries, type of delivery, and number of antenatal clinic visit(s) as confounders in the regression model. The outcome will be fitted first using a two-level bivariate model. Variables found to be significant during the two-level bivariate analysis will be further analyzed using the multinomial regression model (tier 1, tier, and tier 3 categories).

ELIGIBILITY:
1. Inclusion Criteria

   1. Prenatal women in their late pregnancy (near term, term, and post-term pregnancy)
   2. Women who will be in the postpartum time at the endline questionnaire
   3. Women who will live in the selected address for 1 year after delivery
2. Exclusion Criteria

   1. Clients who are in unstable medical states and who are unable to converse without assistance
   2. Women whose postpartum time will be above 1 year at the endline questionnaire
   3. Women who are not available at the selected address for the next 1 year for the endline questionnaire

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Prenatal and postnatal women (females) who found in the selected Kebeles will be included in the study.
Enrollment: 598 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Magnitude (percentage) of postnatal women who use any contraceptive method; 2. The percentage of each contraceptive method (choices) utilized by postnatal women | Recruitment to end of the study: 1 year
  Based on the data obtained from a quantitative questionnaire filled out by each participant, the magnitude of postpartum contraception among postnatal women will be determined at the baseline questionnaire (T0) and at the endline questionnaire (12 months later). Use will be dichotomized into the use of any method versus nothing used. The survey question will be: Do participants currently using any method on a regular basis to space between pregnancies? If they do, then the investigator will pass on to the second question on the method choices. Women's contraceptive preferences for intervention and control populations will be collected at the mentioned time points. Preferences will be dichotomized into more effective and less effective methods. Choices will also be grouped by tiers based on their effectiveness (tier 1, tier 2, and tier 3). The effect of group vs. individual counseling on the use of and preferences for postpartum contraception will then be assessed by using odds ratios.

CONTACTS AND LOCATIONS:
Overall Officials: Zewdie Aderaw Alemu, PhD, Study Director — St. Paul's Hospital Millennium Medical College, Ethiopia
Locations (1):
- St. Paul's Hospital Millennium Medical College, Ethiopia, Addis Ababa, Ethiopia

IPD SHARING:
Plan to Share IPD: Yes
Information can be shared based on request.
Supporting Information: Study Protocol
Time Frame: Currently available